CLINICAL TRIAL: NCT05883085
Title: A Study on the Safety and Effectiveness of Anlotinib for Neoadjuvant Treatment of Locally Advanced, or Unresectable Pheochromocytoma or Paraganglioma
Brief Title: A Study on the Safety and Effectiveness of Anlotinib for Neoadjuvant Treatment of PPGL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06086-02
Record Dates: First submitted 2023-04-10; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-04

CONDITIONS: Pheochromocytoma; Paraganglioma
Keywords: Pheochromocytoma or Paraganglioma; Neoadjuvant Treatment; Anlotinib
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib hydrochloride (Other): Patients receive anlotinib hydrochloride 8-12mg orally once daily on days 1-14. Courses repeat every 21 days
  Interventions: Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Patients receive anlotinib hydrochloride 8-12mg orally once daily on days 1-14. Courses repeat every 21 days
  Other Names: Anlotinib

SUMMARY:
This phase II trial studies the effectiveness of anlotinib hydrochloride in the neoadjuvant therapy of locally advanced, or unresectable pheochromocytoma or paragangliom(PPGL). Anrotinib is used preoperatively in order to change unresectable tumors to resectable and reduce the high risk of surgery.

DETAILED DESCRIPTION:
This prospective, single arm phase II study is designed to evaluate the efficacy of neoadjuvant therapy with anlotinib hydrochloride in locally advanced,or unresectable PPGL patients. Locally advanced,or unresectable PPGL patients receive anlotinib hydrochloride(10-12mg orally once daily on days 1-14, courses repeat every 21 days). Imaging examinations will be conducted after 4 courses to re-evaluate the surgical possibility. If the patient's tumor shrinks after 4 courses but is still unresectable, the patients will continue antirotinib therapy for another 4 courses.

PRIMARY OBJECTIVES:

The proportion of patients whose PPGL change from unresectable to resectable tumor.

SECONDARY OBJECTIVES:

To determine the objective response rate (ORR) . To determine the ratio of tumor shrinkage. To determine the biochemical response . To determine the R0 resection rate. To determine the Major pathological response rate (MPR). To determine the pathologic complete remission（pCR). To assess the safety of anlotinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* The patient is diagnosed as pheochromocytoma or paraganglioma which is unresectable with R0 surgery, or extensive and thus maybe requiring resection of important organs, or with very high surgical risk.
* Laboratory requirements:

  * Absolute granulocyte count (AGC) greater than 1.5 x 109/L;
  * Platelet count greater than 80 x 109/L;
  * Hemoglobin greater than 90g/L;
  * Serum bilirubin less than 1.5 x upper limit of normal (ULN);
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x ULN;
  * Serum creatinine less than 1.5 x ULN or creatinine clearance (CCr)≥60ml/min;
  * Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).
* Confirmed non-pregnancy and lactation. During the entire study period and within 6 months after the last administration, the subjects and their spouses are willing to use efficient contraceptive measures.

Exclusion Criteria:

* Patients who have previously used other anti-vascular targeted drugs, such as sunitinib, bevacizumab, endurance, etc.
* Chemotherapy/systemic therapy, radiotherapy, immunotherapy or surgery within 4 weeks prior to kinase inhibitor therapy.
* Patients with another primary malignancy within 5 years prior to starting study drug.
* Those who have multiple factors that affect oral medications (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.).
* Active or uncontrolled intercurrent illness including, but not limited to:

  * Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg);
  * Patients with uncontrolled myocardial ischemia or myocardial infarction, arrhythmia (including QTC≥480ms), and uncontrolled congestive heart failure，grade ≥2（New York Heart Association ）;
  * Ongoing or active infection;
  * Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment;
  * Renal failure requires hemodialysis or peritoneal dialysis;
  * Have a history of immunodeficiency, including HIV or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
  * Diabetes is poorly controlled (fasting blood glucose (FBG)> 10mmol/L);
  * Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein content is confirmed to be greater than 1.0 g;
* Patients who have seizures and need treatment;
* Any of the following conditions ≤ 6 months prior to registration: Cerebrovascular accident (CVA) or transient ischemic attack (TIA); Serious or unstable cardiac arrhythmia; Pulmonary embolism, untreated deep venous thrombosis (DVT).
* Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders.
* Imaging shows that the tumor has invaded important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study.
* Regardless of the severity, patients with any signs of bleeding or medical history; within 4 weeks before enrollment, patients with any bleeding or bleeding event ≥ CTCAE grade 3, unhealed wounds, ulcers or fractures.
* Participated in other clinical trials within 4 weeks.
* Patients are using drugs that interact with anlotinib.
* Any of the following: Pregnant women, Nursing women, Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Patients with stable disease, and no desire for surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of PPGL patients whose tumor change from unresectable to resectable tumor. | At the end of Cycle 4 (each cycle is 21 days)
  The proportion of PPGL patients whose tumor change from unresectable to resectable

SECONDARY OUTCOMES:
The objective response rate (ORR) | At the end of Cycle 4 (each cycle is 21 days)
  Determined by the RECIST 1.1 criteria
The ratio of tumor shrinkage | At the end of Cycle 4 (each cycle is 21 days)
  The proportion of decrease in the sum of total size of the target lesions after treatment compared to before treatment.
The biochemical response. | At the end of Cycle 4 (each cycle is 21 days)
  An effective response of 24hCA, MNs meant that the concentration decreaseed by more than 40% than the baseline value or decreaseed to the normal range.
R0 resection rate. | At the end of Cycle 4 (each cycle is 21 days)
  The proportion of patients with surgical resection reached R0 resection
Major pathological response rate (MPR). | At the end of Cycle 4 (each cycle is 21 days)
  Defined as the remaining surviving tumor after surgical resection do not exceed 10% of the initial tumor tissue.
Pathologic complete remission (pCR). | At the end of Cycle 4 (each cycle is 21 days)
  There is no tumor cells microscopically.
Safety of anlotinib treatment. | At the end of Cycle 1 (each cycle is 21 days)
  Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Anli Tong, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China